CLINICAL TRIAL: NCT00802087
Title: A Single-Centre, Single Dose, Randomized,Open Label, Exploratory, 5-way Crossover Study Evaluating the Pharmakokinetic Profiles of Various Egalet® Hydrocodone Formulations In Healthy Volunteers Under Fasting Conditions.
Brief Title: Single Dose Pharmacokinetics of Egalet® Hydrocodone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HC-EG-001
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Hydrocodone; Pharmacokinetics; Safety & Tolerability
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Egalet® hydrocodone treatment A (Experimental): Single Dose administration
  Interventions: Drug: hydrocodone
- Egalet® hydrocodone Treatment B (Experimental): Single Dose Administration
  Interventions: Drug: hydrocodone
- Egalet® hydrocodone Treatment C (Experimental): Single Dose Administration
  Interventions: Drug: hydrocodone
- Egalet® hydrocodone Treatment D (Experimental): Single Dose Administration
  Interventions: Drug: hydrocodone
- Active Comparator (Active Comparator): Single Dose Administration
  Interventions: Drug: hydrocodone & acetaminophen combination

INTERVENTIONS:
Drug: hydrocodone — Extended Release tablet
  Arms: Egalet® hydrocodone Treatment B; Egalet® hydrocodone Treatment C; Egalet® hydrocodone Treatment D; Egalet® hydrocodone treatment A
Drug: hydrocodone & acetaminophen combination — Immediate Release tablet, hydrocodone and acetaminophen combination product
  Arms: Active Comparator

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetic profile of different Egalet® hydrocodone formulations and compare to a marketed hydrocodone drug.

DETAILED DESCRIPTION:
Outcomes:

Pharmacokinetic parameters and bioequivalence testing.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* ≥18 and ≤55 years of age
* BMI ≥19 and ≤30.0

Exclusion Criteria:

* Clinically significant abnormalities, physical or psychological illnesses or conditions contraindicating hydrocodone treatment
* History of significant abuse, dependance or addiction of alcohol, drugs or hard drugs within one year prior to screening
* Allergic to hydrocodone, hydromorphone, other opioids, or related drugs
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to study drug administration
* Pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the Pharmacokinetics of Egalet® hydrocodone formulations. PK Parameters: AUC0-t, AUC0-inf, Cmax, Residual Area, Tmax, T½ el, Kel, MRT, proportion of AUC before Tmax, AUC0-12 and AUC0-24 | Single-dose evaluation

SECONDARY OUTCOMES:
To evaluate safety and tolerability of Egalet® hydrocodone formulations. Hematology, biochemistry, urinalysis, ECG, vital signs (including pulse oximetry), and adverse events monitoring. | Single-dose evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christine Andersen, M.Sc.Pharm, Study Director — Egalet A/S
Locations (1):
- Montreal, Quebec, Canada